CLINICAL TRIAL: NCT03330236
Title: Effect of Spectral Edge Frequency and Patient State Index (Electroencephalography) - Guided Anesthetic Care on Delirium After Laparoscopic Surgery: the EMODIPOD Randomized Controlled Trial
Brief Title: EEG - Guided Anesthetic Care and Postoperative Delirium
Acronym: EMODIPOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201612631
Record Dates: First submitted 2017-10-19; First posted 2017-11-06 (Actual); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Delirium; Emergence Delirium; Anesthesia, General; Electroencephalography; Laparoscopy; Surgical Procedures, Operative
Keywords: Electroencephalography; Spectral edge frequency; Patient state index; Anesthesia; Laparoscopic surgery; Postoperative delirium; Emergence delirium
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Intervention Model Description: The study is a prospective, pragmatic, patient and outcome assessor blinded, randomized 1:1 and controlled parallel trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, care providers (excluding the anesthesia team taking care of the patient in the operative room), and outcome assessors are blinded to the results of randomization or group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study arm (Experimental): All patients in the study arm will receive the anesthetic care guided by the SedLine EEG Brain Function Monitor in addition to the conventional monitors. In addition to the conventional/standard interventions of anesthetic care, an additional intervention related to this trial is the anesthetic "depth" management via the titration of the propofol and remifentanil infusion rates to maintain SEF and PSI in the targeted ranges based on the SedLine EEG monitoring.
  Interventions: Device: Anesthetic "depth" management
- Control arm (No Intervention): All patients in the control arm will receive the anesthetic care guided by the conventional monitors only. Patients in the control arm will be monitored using the SedLine EEG Brain Function Monitor; however, the screen of this monitor will be covered by an opaque cloth and blinded to the anesthesia team.

INTERVENTIONS:
Device: Anesthetic "depth" management — The propofol and remifentanil infusion rates will be adjusted to maintain the spectral edge frequency (SEF) value at 10-15 and the patient state index (PSI) value at 25-50 based on the SedLine EEG Brain Function Monitoring.
  Arms: Study arm

SUMMARY:
The study is a prospective, double blinded, randomized and controlled parallel trial to investigate the effect of the anesthetic care guided by EEG monitor (SedLine) on postoperative delirium. EMODIPOD = Electroencephalography Monitoring tO Decrease the Incidence of PostOperative Delirium

DETAILED DESCRIPTION:
To investigate the impact of the anesthetic care guided by EEG monitor (SedLine) on (1) the incidence of delirium in post-anesthesia care unit (PACU) and within the first five days after laparoscopic surgery and (2) the incidence of in-hospital complications and 30-day mortality in adult patients after laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years;
2. ASA Physical Score I-III
3. Scheduled to undergo elective laparoscopic surgeries under general anesthesia with endotracheal intubation;
4. Extubation expected after surgery;
5. Scheduled to stay in hospital for > 3 days after surgery.

Exclusion Criteria:

1. Refuse to participate;
2. Emergent surgery;
3. Trauma patients;
4. Preoperative cognitive impairment characterized by Mini-Mental State Examination (MMSE) of 23 or less;
5. Preoperative history of stroke, schizophrenia, major depression, Parkinson's disease, epilepsy, or dementia;
6. Inability to communicate in the preoperative period due to illiteracy, language difficulties, or significant hearing or visual impairment;
7. Inability to complete MMSE and delirium survey;
8. Severe cardiac disease including low-output cardiac failure defined as a preoperative left ventricular ejection fraction < 30%, or arrhythmia with pacemaker or AICD placement;
9. Severe hepatic dysfunction being evaluated for liver transplantation or with a Child- Pugh Class C classification;
10. Severe renal dysfunction requiring renal replacement therapy before surgery;
11. Those with preoperative ASA classification of 4 or who are unlikely to survive for more than 3 days after surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Stavris, Study Director — Yale School of Medicine Department of Anesthesiology
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 70,783 patients scheduled to undergo an elective surgical procedure in the main operating rooms at Xiangya Hospital from October 2017 to August 2019, a total of 1,560 participated in this study.
Groups:
- EEG Guided: All patients in the EEG Guided study arm will receive the anesthetic care guided by the SedLine EEG Brain Function Monitor in addition to the conventional monitors. In addition to the conventional/standard interventions of anesthetic care, an additional intervention related to this trial is the anesthetic "depth" management via the titration of the propofol and remifentanil infusion rates to maintain SEF and PSI in the targeted ranges based on the SedLine EEG monitoring.
  Anesthetic "depth" management: The propofol and remifentanil infusion rates will be adjusted to maintain the spectral edge frequency (SEF) value at 10-15 and the patient state index (PSI) value at 25-50 based on the SedLine EEG Brain Function Monitoring.
- Usual Care: All patients in the usual care arm (control) will receive the anesthetic care guided by the conventional monitors only. Patients in the control arm will be monitored using the SedLine EEG Brain Function Monitor; however, the screen of this monitor will be covered by an opaque cloth and blinded to the anesthesia team.
Period: Overall Study
Arm/Group | EEG Guided | Usual Care
Started | 779 | 781
Received Surgery | 779 | 781
Modified ITT (Participants analyzed as the Modified ITT analysis population.) | 773 | 774
Completed | 679 | 697
Not Completed | 100 | 84
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 4 | 3
Not completed — SedLine malfunction/blinding | 19 | 14
Not completed — Volatile anesthetics used | 11 | 8
Not completed — Surgery aborted/converted to open | 60 | 52

BASELINE CHARACTERISTICS:
Population: Modified ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | EEG Guided | Usual Care | Total
Number analyzed (Participants) | 773 | 774 | 1547
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [55 to 67] | 61 [55 to 67] | 61 [55 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335 | 315 | 650
  Male | 438 | 459 | 897
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 773 | 774 | 1547
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 773 | 774 | 1547

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Delirium
Description: The Number of Participants with Postoperative Delirium is operationally defined as the count of patients with postoperative delirium. Postoperative delirium is an acute brain dysfunction characterized by inattention, disorganized thinking, and a fluctuating course.
Time Frame: up to five (5) days after surgery
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 773 | 774
Participants | 8 | 9

2. Secondary Outcome: Emergence Delirium
Description: Incidence (count) of emergence delirium at post-anesthesia care unit (PACU)
Time Frame: 30 min following the extubation
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 773 | 774
Participants | 91 | 102

3. Secondary Outcome: Non-delirium Complications
Description: Complications after surgery such as acute kidney injury, cardiac events, cerebrovascular events, renal injury, GI complications, infections (etc) were assessed using the Clavien-Dindo classification. Reported are the count of those with a composite complication Clavien-Dindo Grade ≥II.
  The classifications are as follows:
  Grade I = Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.
  Grade II = Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusionsand total parenteral nutritionare also included.
  Grade III = Requiring surgical, endoscopic or radiological intervention; IIIa = Intervention not under general anesthesia; IIIb = Intervention under general anesthesia.
  Grade IV = Life-threatening complication (including CNS complications)* requiring IC/ICU-management; IVa = single organ dysfunction (including dialysis); IVb
Time Frame: within 30 days after surgery
Population: Modified ITT population/patients with valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 768 | 773
Participants | 175 | 193

4. Secondary Outcome: GI Functional Recovery
Description: Speed of GI functional recovery (pass gas)
Time Frame: within 30 days after surgery
Population: These data were not collected and analyzed.
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: All-cause 30-day Mortality
Description: All-cause 30-day mortality
Time Frame: 30 days after surgery
Population: Modified ITT population/patients with complete data
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 765 | 767
Participants | 2 | 1

6. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay was counted from the day of surgery (day 0) to the day when the patient was ready for discharge.
Time Frame: up to 30 days after surgery
Population: Modified ITT population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 773 | 774
days | 6 [3 to 8] | 6 [3 to 8]

7. Secondary Outcome: ICU Admission
Description: Count of patients that were admitted to ICU after surgery.
Time Frame: up to 72 hours
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 773 | 774
Participants | 17 | 15

8. Secondary Outcome: Length of ICU Stay
Description: the duration of time when the patient residing in ICU
Time Frame: up to 30 days after surgery
Population: These data were not collected and analyzed.
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: NRS Pain Score
Description: Numeric Rating Scale subjective pain where 0 indicates no pain and 10 indicates the worst pain.
Time Frame: 24 hours after surgery
Population: These data were not collected and analyzed.
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: NRS Sleep Score
Description: Numeric Rating Scale subjective sleep quality at 8:00 am where 0 indicates best possible sleep and 10 indicates worst possible sleep
Time Frame: 24 hours after surgery
Population: These data were not collected and analyzed.
Arm/Group | EEG Guided | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days post surgery
Arm/Group | EEG Guided | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/779 | 1/781
Serious Adverse Events (participants affected / at risk) | 0/779 | 0/781
Other Adverse Events (participants affected / at risk) | 3/779 | 3/781
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EEG Guided (N=779) | Usual Care (N=781)
Intraoperative awareness (General disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03330236/Prot_SAP_000.pdf